CLINICAL TRIAL: NCT04714814
Title: a Multi-omics Cohort Study of Mechanisms of Fate Evolution of Colorectal Adenocarcinoma Metastasis
Brief Title: Mechanisms of Fate Evolution of Colorectal Adenocarcinoma Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government); RenJi Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Metastatic CRC cell fate
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer Stage III; Colorectal Cancer Stage IV
Keywords: Colorectal , Metastatisis ,Cancer Cell Fate Regulatory Mechanism
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue samples, blood samples, stool, pleural effusion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a two stage nested case-control study to construct the hologram plane , explore biomarkers and screening original drugs of metastatic colorectal cancer.

DETAILED DESCRIPTION:
Stage Ⅰ is a cross-sectional study to record selected information and biospecimen of more than 200 colorectal cancer cases( at least 160 stage Ⅲ cases,40 stage Ⅳ（synchronous metastasis）).Stage Ⅱ is a nested case-control study. 200 eligible cases enrolled in phaseⅠwill be followed up for 5 years to record recurrence, metastasis and to collect biospecimen . Each case with the study outcome will be matched with the corresponding control according to the proportion of 1:1 according to age, sex and other conditions, and further analysis will be made.

ELIGIBILITY:
Inclusion Criteria:

* Baseline population (stage III colorectal cancer) inclusion criteria:

  1. Aged 18-75.
  2. Physical condition (ECOG) score ≤ 1.
  3. Colorectal adenocarcinoma was confirmed by histopathology.
  4. No family history of hereditary tumor.
  5. Accept standard radical resection of colorectal cancer, R0 resection, number of lymph node dissection ≥ 12.
  6. Preoperative clinical stage is stage III.
  7. Agree to receive standard fluorouracil ±oxaliplatin adjuvant chemotherapy for 3 to 6 months.
  8. Enough primary surgical or biopsy tissues for examination.
  9. Enough peripheral blood samples for examination.
  10. Agree to sign informed consent to participate in this project.

Baseline population (stage Ⅳ colorectal cancer) inclusion criteria:

1. Aged 18-75.
2. Histopathological diagnosed colonic or rectal adenocarcinoma of stage IV.
3. Not yet received antineoplastic therapy.
4. Baseline imaging evaluation shows at least one measurable focus.
5. Sufficient primary surgical or biopsy tissues and metastatic tissues of at least one organ for examination.
6. Enough peripheral blood samples for examination.
7. Expected survival time ≥ 3 months.
8. Provide information such as demography, current medical history or current tumor disease, pathological diagnosis and staging of tumor, physical status of ECOG, radiographic evaluation of tumor, etc.
9. Agree to sign informed consent to participate in this project.

Metastasis colorectal cancer cohort study inclusion criteria:

1. Aged 18-75.
2. Physical condition (ECOG) score ≤ 1.
3. Colorectal adenocarcinoma was confirmed by histopathology.
4. No family history of hereditary tumor.
5. Accept standard radical resection of colorectal cancer, R0 resection, number of lymph node dissection ≥ 12.
6. Preoperative clinical stage is stage III and the postoperative pathological stage was confirmed as stage III.
7. Agreed to receive standard fluorouracil ±oxaliplatin adjuvant chemotherapy for 3 to 6 months.
8. Enough primary surgical or biopsy tissues for examination.
9. Enough peripheral blood samples for examination.
10. Agree to sign informed consent to participate in this project.

Exclusion Criteria:

* Baseline population (stage III colorectal cancer) exclusion criteria:

  1. Participating in interventional clinical studies or receiving research treatments that influence patients' treatment decisions.
  2. Postoperative pathological stage was confirmed as stage II.
  3. Abnormal function of heart, lung, liver, kidney, hematopoiesis or bone marrow reserve, which cannot tolerate operation or chemotherapy.
  4. Diagnosed with malignant tumors that have progressed or need to be treated in the past 5 years, except for cured skin basal cells and skin squamous cell carcinoma.
  5. Having mental illness or other serious cardiovascular diseases.
  6. Pregnancy or lactation or planned pregnancy within one year.
  7. Emergency operation (perforation, bleeding, intestinal obstruction, etc.).

Baseline population (stage Ⅳcolorectal cancer) exclusion criteria:

1. Family history of hereditary colorectal cancer, such as Lynch syndrome, familial adenomatous polyposis, P-J syndrome, etc.
2. Nervous system metastasis.
3. Complicated with other malignant tumors.
4. Having poorly controlled chronic concomitant diseases that affect the prognosis.
5. Any complication that may affect the results of the study .

Metastasis colorectal cancer cohort study exclusion criteria:

1. Participating in interventional clinical studies or receiving research treatments that influence patients' treatment decisions.
2. Abnormal function of heart, lung, liver, kidney, hematopoiesis and bone marrow reserve, which cannot tolerate operation and chemotherapy.
3. Diagnoses with malignant tumors that have progressed or need to be treated in the past 5 years, except for cured skin basal cells and skin squamous cell carcinoma.
4. Having mental illness or other serious cardiovascular disease.
5. Pregnancy or lactation or planned pregnancy within one year.
6. Emergency operation (perforation, bleeding, intestinal obstruction, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with CRC (Stage III and Stage IV)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
recurrence or metastasis provened by imageologic diagnosis (PFS) | May 31, 2023
  tumor metastasis or progression occurred during the enrolment period

CONTACTS AND LOCATIONS:
Overall Officials: Sun Jing, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ruijin Hospttal, Shanghai, Sahgnhai, China